CLINICAL TRIAL: NCT04923984
Title: Embolization of Middle Meningeal Artery for Subdural Hematoma in Canada -EMMA-Can
Brief Title: Embolization of Middle Meningeal Artery for Subdural Hematoma in Canada (EMMA Can)
Acronym: EMMA-Can
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Jai Shankar, Professor, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HS24152(B2020-077)
Record Dates: First submitted 2021-06-07; First posted 2021-06-11 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Subdural Hematoma
Keywords: Embolization; Middle Meningeal Artery; Chronic Subdural Hematoma
MeSH Terms: conditions — Hematoma, Subdural; Hematoma, Subdural, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Embolization of Middle Meningeal Artery for Subdural Hematoma (Experimental): All patients with CSDH will undergo embolization of Middle Meningeal artery
  Interventions: Procedure: Embolization of the middle meningeal artery

INTERVENTIONS:
Procedure: Embolization of the middle meningeal artery — embolization of the middle meningeal artery with an embolic agent (Microparticles, liquid embolic agents, SwiftPAC coils or others).

SUMMARY:
EMMA-Can is a prospective cohort study to assess the safety and effectiveness of MMA-embolization for the treatment of CSDH.

Hypothesis- EMMA reduces the recurrence rate of CSDH with or without concomitant surgical evacuation.

DETAILED DESCRIPTION:
The purpose of our study is to conduct a prospective cohort study to assess the safety and effectiveness of MMA embolization for the treatment of CSDH. All patients with CSDH presenting to the emergency room or to neurosurgical outpatient clinic will be screened for potential enrollment. If the subject is willing to participate an informed consent will be obtained.

All patients presenting to the emergency room or in neurosurgery clinic with CSDH diagnosed on CT scan will be considered for the study. If the patient needs emergent evacuation for clinical reasons, patient will be taken for surgical evacuation before consideration of EMMA. Patients that are more likely to have recurrence after surgical evacuation are those with recurrent CSDH, on antiplatelet or antithrombotic treatment. The EMMA could be used as primary treatment or in conjunction with surgery in these patients or in patients who may not be good surgical candidate.

Follow up - All patients will be followed after discharge from the hospital at 1, 3, 6 and 12 months interval. The follow up at 3 months will include plain CT head of the patient, which is standard of care for most patients. The follow up at 6 and 12 months will be only clinical follow up.

Patients will be assessed for recurrence of CSDH on CT scan of head. Symptoms associated with the recurrence will be recorded. The size of the CSDH will be measured and compared to previous scans and peri-procedural morbidity and mortality related to EMMA will be sought. This will be done at 3 months post EMMA.

ELIGIBILITY:
Inclusion Criteria:

- All patients with subdural hematoma coming to the emergency room or to neurosurgical outpatient clinic.

Exclusion Criteria:

* If informed consent cannot be obtained from the patient or their substitute decision maker.
* Known allergy to liquid embolic agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Radiographic recurrence | up to 90-days for EMMA
  Recurrence of CSDH on imaging (CT scan or MRI) of head .
Symptomatic recurrence | up to 90-days from EMMA
  Symptomatic recurrence attributable to the side of the CSDH on imaging (CT scan or MRI) of head

SECONDARY OUTCOMES:
Size | 30 days and 90 days
  Change in size of the CSDH
Mortality within 90-days | up to 90-days
  Peri-procedural mortality related to EMMA.
90 day Modified Rankin Score </=3 | 90-days
  Percentage of patients with a Modified Rankin score </=3
Reduction of CSDH size at 90-days | 90-days
  Reduction of the size of the CSDH on CT scan of the head at 90-days from EMMA
Morbidity within 90-days | up to 90-days
  peri-procedural morbidity related to EMMA such as puncture site hematoma, arterial dissection or stroke
90-day MOCA and EQ-5D-5L health score | Day 90
  score on the Montreal Cognitive Assessment test and score on the EQ-5D-5L assessment
Discharge destination | up to 100 weeks
  discharge location from acute care
Length of hospital stay | up to 100 weeks
  number of days of acute care hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Jai Shankar, MD, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences centre, Winnipeg MB, Manitoba, Canada